CLINICAL TRIAL: NCT07138534
Title: Investigation of the Effect of Prehabilitation Practice on Patient Outcomes in Frail Patients Planned for Elective Coronary Artery Bypass Graft
Acronym: ERAS
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bahçeşehir University (Other)
Responsible Party: Principal Investigator, Gamze ataman YILDIZ, Surgical Nurse, Bahçeşehir University
Allocation: Randomized | Model: Sequential | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 20250715
Record Dates: First submitted 2025-08-05; First posted 2025-08-24 (Actual); Last update posted 2025-08-24 (Actual); Status verified 2025-08

CONDITIONS: Coronary Artery Bypass Graft (CABG)
Keywords: frail patients; coronary artery bypass
MeSH Terms: interventions — Preoperative Exercise

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- routine procedure (No Intervention): control
- prehabilitation (Experimental): In addition to exercise programmes, it includes nutritional optimisation, psychosocial preparation and smoking cessation.
  Interventions: Behavioral: prehabilitation

INTERVENTIONS:
Behavioral: prehabilitation — In addition to exercise programmes, it includes nutritional optimisation, psychosocial preparation and smoking cessation.
  Arms: prehabilitation

SUMMARY:
The basic concept of prehabilitation is to increase the functional capacity of the individual to withstand an expected injury. It embodies the idea of being proactive against the common reactive approach of rehabilitation. While the initial prehabilitation model was limited to physical training, it has now evolved into a multimodal entity that includes nutritional optimisation, psychosocial preparation and smoking cessation in addition to exercise programmes. In the last decade, there has been an increasing effort to coincide prehabilitation with surgery, as surgery is rightly perceived as a stressor for human structural and physiological functions.

DETAILED DESCRIPTION:
Frailty is an increasingly recognised risk factor for surgery. The degree of frailty and how this may affect postoperative recovery profiles is unclear. Preoperative frailty may predispose patients to worse outcomes in cardiac surgery; however, there is limited data on how preoperative frailty affects patient outcomes through prehabilitation practices.

ELIGIBILITY:
Inclusion Criteria:

* frail patient

Exclusion Criteria:

* frail patient

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
patients' activities of daily living | It will be measured one month after the surgery. The date may vary depending on the patient.
  Patients' daily living activities will be assessed according to the Katz Daily Living Activities Scale. Those with high scores will be shown to have better daily living activities. scale name: Katz activities of daily living. 6 is the highest score and 0 is the lowest. A score of 6 means completely independent.
functional capacity | It will be evaluated one month after surgery. The date may vary depending on the patient.
  Patients' functional capacities will be assessed using the Duke Activity Scale. Those with high scores will be confirmed to have better physical and functional capacities. scale name: Duke Activity Status Index. The lowest score is 0 and the highest score is 58.2. A score of 58.2 indicates the highest functional capacity.
Nutritional Status | It will be evaluated one month after surgery. The date may vary depending on the patient.
  Patients' nutrition will be assessed using a mini nutritional test. Those who score high will be assumed to be in good nutritional condition. scale name: Mini nutritional test. The highest score is 14 and the lowest is 0. The highest score indicates the absence of malnutrition.
Post-operative recovery status | It will be measured one month after the surgery.
  The patient's physical, psychological, bowel activity and general condition will be assessed using a post-operative recovery index. Those with high scores will be considered to have recovered better. The scale name is the postoperative recovery index. The index consists of 5 sub-dimensions and 25 items. The sub-dimensions are psychological symptoms, physical activities, and general symptoms. The ASII total and sub-dimension scores are bowel symptoms and desire-urge symptoms. When determining the subscale score, the scores of the relevant items are summed and the arithmetic mean is calculated. For the total score, all items are summed and the arithmetic mean is calculated. High scores on the index indicate greater difficulty in post-operative recovery, while low scores indicate that post-operative recovery is easier. The ASII is a reliable and valid tool for assessing

CONTACTS AND LOCATIONS:
Overall Officials: FATMA ETİ ASLAN, Proffesor, Study Director — Bahcesehir Universty

IPD SHARING:
Plan to Share IPD: No
The study has not yet begun, so we do not know at this point whether there will be any objections to sharing the data once it has been collected. Therefore, we can say that it will not be shared at this time.

REFERENCES:
- [Background] Steinmetz C, Bjarnason-Wehrens B, Walther T, Schaffland TF, Walther C. Efficacy of Prehabilitation Before Cardiac Surgery: A Systematic Review and Meta-analysis. Am J Phys Med Rehabil. 2023 Apr 1;102(4):323-330. doi: 10.1097/PHM.0000000000002097. Epub 2022 Sep 23. PMID 36149383
- See also: This page is related to Eras cardiac. It is a recommendation from the Eras prehabilitation guidelines. This study was deemed appropriate due to the very low level of evidence. — https://www.erascardiac.org/

DOCUMENTS (2):
  • Study Protocol (2024-03-11): https://cdn.clinicaltrials.gov/large-docs/34/NCT07138534/Prot_000.pdf
  • Informed Consent Form (2019-01-02): https://cdn.clinicaltrials.gov/large-docs/34/NCT07138534/ICF_001.pdf